CLINICAL TRIAL: NCT06189924
Title: Proteomic Analysis of Exhaled Breath Condensate in Mechanically Ventilated Intensive Care Patients
Brief Title: Exhaled Breath Condensate Analysis in Mechanically Ventilated Patients
Status: Not yet recruiting | Type: Observational
Sponsor: The Institute of Molecular and Translational Medicine, Czech Republic (Other)
Responsible Party: Sponsor
Other Study IDs: 64734
Record Dates: First submitted 2023-12-04; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Acute Respiratory Failure; Critical Illness
Keywords: exhaled breath condensate; proteomics; genomics; mechanical ventilation; acute respiratory failure; lung injury; intensive care
MeSH Terms: conditions — Critical Illness; Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mechanically ventilated patients with primary or secondary lung injury: Mechanically ventilated patients with primary or secondary lung injury due to various pathologies. Patients will be treated at intensive care units (ICU).
  Interventions: Diagnostic Test: Proteomic analysis of exhaled breath condensate
- Mechanically ventilated patients without lung injury: Mechanically ventilated patients without lung injury, with various pathologies. Patients will be treated at intensive care units (ICU).
  Interventions: Diagnostic Test: Proteomic analysis of exhaled breath condensate

INTERVENTIONS:
Diagnostic Test: Proteomic analysis of exhaled breath condensate — Mechanically ventilated intensive care patients will be sampled for exhaled breath condensate from the ventilator circuit.
  Other Names: Molecular biological examination of the venous blood sample

SUMMARY:
Mechanically ventilated intensive care patients will be sampled for a small amount of exhaled breath condensate from the ventilator circuit and for venous blood.

Proteomic analysis of the exhaled breath condensate will be performed using mass spectrometry and in the blood sample, corresponding changes in the DNA, RNA, proteins, and metabolites will be studied. Resulting profiles will be correlated with routinely monitored parameters in order to identify patterns corresponding to various pathologies in order to enable their early detection.

DETAILED DESCRIPTION:
Exhaled breath condensate (EBC) is a product of gas exchange in the lungs. It contains plethora of substances of possible diagnostic value and its composition is likely to change rapidly in response to the development of pathological conditions, especially in the lungs.

Mechanically ventilated intensive care patients with various pathological conditions will be sampled for a small amount of EBC from the ventilator circuit and for venous blood. A sampling method not affecting relevant parameters of mechanical ventilation will be developed and standardised.

EBC samples will be frozen and after processing, proteomic analyses will be performed using mass spectrometry. In the blood sample, corresponding changes in the DNA, RNA, proteins, and metabolites will be studied using molecular biological methods. Resulting profiles will be correlated with routinely monitored parameters (such as inflammation markers, microbiological findings and mechanical ventilation parameters) with the aim of finding patterns corresponding to the early stages of various pathological conditions focusing on lung tissue. Identification of patterns specific to initial stages of lung and other organ pathologies would enable their early treatment possibly shortening mechanical ventilation/ICU stay and reducing morbidity/mortality.

ELIGIBILITY:
Inclusion Criteria:

Intensive care setting Mechanical ventilation Ventilator/ventilator circuit technically suitable for sampling of exhaled breath condensate

Exclusion Criteria:

Mechanical ventilation challenging to the extent that the insertion of the sampling kit into the ventilator circuit would substantially increase the risk for respiratory deterioration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated intensive care patients with or without acute hypoxemic respiratory failure
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of proteomic patterns of the exhaled breath condensate in mechanically ventilated intensive care patients. | January 2024 - December 2029
  Proteomic patterns of the exhaled breath condensate will be studied in mechanically ventilated intensive care patients. The results will be analysed and compared with the aim to identify patterns specific for the pathological conditions.

SECONDARY OUTCOMES:
Correlation of exhaled breath condensate patterns with molecular biological findings in venous blood - DNA | January 2024 - December 2029
  Venous blood sample will be analysed employing targeted analyses of DNA. The results will be correlated to proteomic patterns obtained from the exhaled breath condensate.
Correlation of exhaled breath condensate patterns with molecular biological findings in venous blood - RNA | January 2024 - December 2029
  Venous blood sample will be analysed employing targeted analyses of RNA. The results will be correlated to proteomic patterns obtained from the exhaled breath condensate.
Correlation of exhaled breath condensate patterns with molecular biological findings in venous blood - proteins | January 2024 - December 2029
  Venous blood sample will be analysed employing targeted analyses of proteins. The results will be correlated to proteomic patterns obtained from the exhaled breath condensate.
Correlation of exhaled breath condensate patterns with molecular biological findings in venous blood - metabolites | January 2024 - December 2029
  Venous blood sample will be analysed employing targeted analyses of metabolites. The results will be correlated to proteomic patterns obtained from the exhaled breath condensate.

CONTACTS AND LOCATIONS:
Overall Officials: Emil Berta, MD PhD, Principal Investigator — IMTM, Palacky University in Olomouc, Faculty of Medicine and Dentistry
Locations (2):
- Czechia (2):
  - Institute of Molecular and Translational Medicine, Palacky University, Olomouc
  - University Hospital Olomouc, Olomouc

IPD SHARING:
Plan to Share IPD: Undecided